CLINICAL TRIAL: NCT02274857
Title: Randomized Evaluation of Atrial Fibrillation Treatment With Focal Impulse and Rotor Modulation Guided Procedures (REAFFIRM)
Brief Title: Randomized Evaluation of Atrial Fibrillation Treatment With Focal Impulse and Rotor Modulation Guided Procedures
Acronym: REAFFIRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: REAFFIRM
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Results first posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Focal Impulse and Rotor Modulation Mapping Catheter (FIRMap); Rotor; FIRM-guided procedure; REAFFIRM
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard PVI Ablation (Active Comparator): Standard catheter ablation including pulmonary vein isolation (PVI) procedure for the treatment of persistent AF.
  Interventions: Procedure: Standard PVI Ablation
- FIRM-guided Procedure and PVI (Experimental): FIRM-guided procedure followed by standard catheter ablation including PVI.
  Interventions: Procedure: FIRM-Guided Procedure and PVI

INTERVENTIONS:
Procedure: Standard PVI Ablation — Standard PVI procedure without FIRMap.
  Other Names: Pulmonary vein isolation; Ablation; Arrhythmia; Persistent atrial fibrillation; Mapping
  Arms: Standard PVI Ablation
Procedure: FIRM-Guided Procedure and PVI — FIRM-guided procedure followed by conventional ablation including PVI.
  Other Names: Pulmonary vein isolation; Ablation; Arrhythmia; Persistent atrial fibrillation; Mapping; FIRMap
  Arms: FIRM-guided Procedure and PVI

SUMMARY:
The study is a prospective, multicenter, randomized study to assess the safety and effectiveness of FIRM procedures followed by conventional ablation including PVI versus a standard PVI procedure for the treatment of persistent atrial fibrillation (AF).

ELIGIBILITY:
Key Inclusion Criteria:

* At least two (2) documented episodes of persistent atrial fibrillation during prior 3 months
* Refractory, intolerant, or contraindicated to Class I or III anti-arrhythmic medications
* Left atrial diameter < 6.0 cm

Key Exclusion Criteria:

* Previous AF Ablation
* Presence of structural heart disease
* New York Heart Association (NYHA) Class IV.
* Ejection fraction < 35%.
* History of myocardial infarction (MI) within the past three months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-11-10 (Actual); Study Completion 2018-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Brachmann, MD, Principal Investigator — Klinikum Coburg GmbH
Locations (18):
- United States (10):
  - Arizona Heart Rhythm Center, Phoenix, Arizona
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University - Krannert Institute of Cardiology, Indianapolis, Indiana
  - St. Vincent Hospital, Indianapolis, Indiana
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Hackensack UMC, Hackensack, New Jersey
  - Weill Medical College at Cornell University, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
- Germany (7):
  - Herz- und Diabeteszentrum Bad Oeynhausen, Bad Oeynhausen, Minden-Lübbecke
  - Unfallkrankenhaus Berlin, Berlin
  - Klinikum Coburg GmbH, Coburg
  - Zentrum für klinische Prüfungen in der Facharztzentrum Dresden-Neustadt GbR, Dresden
  - Städtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - Leipzig Heart Institute GmbH, Leipzig
  - Kardiologische Gemeinschaftspraxis am Park Sanssouci, Potsdam
- Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard PVI Ablation: Standard catheter ablation including pulmonary vein isolation (PVI) procedure for the treatment of persistent atrial fibrillation (AF).
  Standard PVI Ablation: Standard PVI procedure without Focal Impulse and Rotor Modulation Mapping Catheter (FIRMap).
- FIRM-guided Procedure and PVI: Focal Impulse and Rotor Modulation (FIRM)-guided procedure followed by standard catheter ablation including PVI.
  FIRM-Guided Procedure and PVI: FIRM-guided procedure followed by conventional ablation including PVI.
Period: Overall Study
Arm/Group | Standard PVI Ablation | FIRM-guided Procedure and PVI
Started | 179 | 171
Completed Per Protocol (Per protocol are subjects in ITT group who completed all follow-ups with no major deviations.) | 102 | 114
Completed | 159 | 165
Not Completed | 20 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 3 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Trial screen failure | 0 | 2
Not completed — Withdrawal by Subject | 11 | 2
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard PVI Ablation | FIRM-guided Procedure and PVI | Total
Number analyzed (Participants) | 179 | 171 | 350
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (8.7) | 64.2 (8.4) | 63.4 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 45 | 97
  Male | 127 | 126 | 253
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 167 | 160 | 327
  Unknown or Not Reported | 8 | 10 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 171 | 159 | 330
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  Netherlands | 27 | 23 | 50
  United States | 80 | 80 | 160
  Germany | 72 | 68 | 140
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.12 (5.63) | 31.17 (5.59) | 31.15 (5.60)
NYHA Classification [Number; unit: category] — The New York Heart Association Functional Classification provides a simple way of classifying the extent of heart failure. It places patients in one of four categories based on how much they are limited during physical activity; the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina.
  Class I = no limitation of physical activity. Class II = slight limitation Class III = marked limitation Class IV = unable to carry on any physical activity without discomfort.
  category
    Class I | 63 | 53 | 116
    Class II | 52 | 63 | 115
    Class III | 18 | 17 | 35
Largest Left Atrial Diameter [Mean (Standard Deviation); unit: mm] | 45.63 (9.63) | 48.07 (7.65) | 46.82 (8.80)
LV Ejection Fraction [Mean (Standard Deviation); unit: %] | 54.5 (8.9) | 53.8 (8.0) | 54.2 (8.5)
Prior and concomitant antiarrhythmic drugs (AAD) [Number; unit: participants] — Prior and concomitant use of AADs refers to the types of pharmacological therapies a participant has been on or is on in order to treat their arrhythmia. Participants may be on more than one type of AAD.
  Class 1 AAD = Sodium Channel Blockers Class 2 AAD = Beta-Adrenoceptor Antagonist Class 3 AAD = Potassium Channel Blockers Class 4 AAD = Calcium Channel Blockers
  participants
    Class I AAD | 29 | 32 | 61
    Class 2 AAD | 115 | 106 | 221
    Class 3 AAD | 67 | 69 | 136
    Class 4 AAD | 21 | 22 | 43
Hospitalizations for Cardiac Arrhythmias within 6 months of screening [Count of Participants; unit: Participants] | 59 | 48 | 107
Treated for atrial fibrillation in the 6 months prior to enrollment [Number; unit: %] | 85.4 | 88.9 | 87.1
History of significant past and/or concomitant diseases or past surgeries [Number; unit: %]
  Cardiovascular | 72.1 | 67.8 | 70.0
  CNS/Neurological | 10.6 | 11.7 | 11.1
  Dermatologic | 5.0 | 4.7 | 4.9
  Drug Allergy | 3.4 | 1.8 | 2.6
  Endocrine/Metabolic | 37.4 | 30.4 | 34.0
  Eyes/Ears/Nose/Throat | 11.2 | 12.9 | 12.0
  Gastrointestinal | 18.4 | 23.4 | 20.9
  Genitourinary | 8.9 | 12.9 | 10.9
  Hematologic | 5.0 | 4.1 | 4.6
  Hepatic | 2.2 | 2.9 | 2.6
  Immunological | 3.9 | 4.7 | 4.3
  Malignancy | 5.6 | 5.3 | 5.4
  Musculoskeletal | 26.3 | 28.1 | 27.1
  Psychiatric | 7.3 | 5.8 | 6.6
  Renal | 8.9 | 11.1 | 10.0
  Respiratory | 24.0 | 22.8 | 23.4
  Other | 21.2 | 26.3 | 23.7
Subjects that had LV Ejection Fraction Measured [Count of Participants; unit: Participants] | 170 | 160 | 330

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Procedure-related Serious Adverse Events (SAEs) Within 7-10 Days of the Procedure
Time Frame: Within 7-10 days of the Procedure
Population: Intent to Treat (ITT) group, defined as subject randomized to a treatment group who had a mapping and/or ablation catheter inserted
Measure: Number; unit: % of participants
Arm/Group | Standard PVI Ablation | FIRM-guided Procedure and PVI
Number analyzed (Participants) | 179 | 171
% of participants | 92.7 | 88.9
Statistical Analysis 1: Comparison: Standard PVI Ablation vs FIRM-guided Procedure and PVI; Test type: Superiority; p = 0.2179, Chi-squared

2. Primary Outcome: Single-procedure Freedom From AF/AT Recurrence at 3 Month Post Index Procedure.
Time Frame: 3-month follow up
Population: ITT: each subject randomized to a treatment group who had a mapping and/or ablation catheter inserted Per Protocol: those subjects in the ITT group who completed all follow-up visits and had no major protocol deviations
Measure: Number; unit: % of participants
Arm/Group | Standard PVI Ablation | FIRM-guided Procedure and PVI
Number analyzed (Participants) | 179 | 171
% of participants | 76.9 | 71.8
Statistical Analysis 1: Comparison: Standard PVI Ablation vs FIRM-guided Procedure and PVI; Test type: Superiority; p = 0.2782, Chi-squared

3. Primary Outcome: Single-procedure Freedom From AF/AT Recurrence at 3 to 12 Months Post Index Procedure.
Time Frame: 3-12 months post study treatment
Population: ITT group, defined as each subject randomized to a treatment group who had a mapping and/or ablation catheter inserted
Measure: Number; unit: % of participants
Arm/Group | Standard PVI Ablation | FIRM-guided Procedure and PVI
Number analyzed (Participants) | 179 | 171
% of participants | 67.5 | 69.3
Statistical Analysis 1: Comparison: Standard PVI Ablation vs FIRM-guided Procedure and PVI; Test type: Superiority; p = 0.7266, Chi-squared

4. Primary Outcome: Freedom From Procedure-related SAEs (Including Those Related to Any Repeat Procedures) Within 12-months of the Initial Procedure
Time Frame: 3 to 12 months post study treatment
Population: ITT group, defined as each subject randomized to a treatment group who had a mapping and/or ablation catheter inserted
Measure: Count of Participants; unit: Participants
Arm/Group | Standard PVI Ablation | FIRM-guided Procedure and PVI
Number analyzed (Participants) | 163 | 167
Participants | 146 | 144
Statistical Analysis 1: Comparison: Standard PVI Ablation vs FIRM-guided Procedure and PVI; Test type: Superiority; p = 0.3522, Chi-squared

5. Secondary Outcome: Evaluate the Acute Effectiveness of FIRM-guided Procedures in Eliminating the Source of Arrhythmia as Shown by: No Evidence of the Source in FIRMap Post-op, OR Reduction of Electrogram Amplitude to < 0.2 Millivolts
Time Frame: Immediately post procedure
Population: ITT
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | FIRM-guided Procedure and PVI
Number analyzed (Participants) | 171
% of participants | 86.1 [79.7 to 91.1]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Standard PVI Ablation | FIRM-guided Procedure and PVI
All-Cause Mortality (participants affected / at risk) | 1/179 | 2/171
Serious Adverse Events (participants affected / at risk) | 19/179 | 28/171
Other Adverse Events (participants affected / at risk) | 0/179 | 0/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard PVI Ablation (N=179) | FIRM-guided Procedure and PVI (N=171)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arteriovenous fistula operation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 3 (5) | 3 (4)
Atrial tachycardia (Cardiac disorders) | 5 (8) | 3 (3)
C-reactive protein increased (General disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 2 (2)
Cerebrovascular accident (Vascular disorders) | 1 (1) | 0 (0)
Fluid overload (Cardiac disorders) | 1 (1) | 1 (1)
Gastroparesis postoperative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 3 (3) | 8 (8)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis infective (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial disease (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial hemmorrhage (Cardiac disorders) | 2 (2) | 0 (0)
Peritoneal hemorrhage (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Vessel puncture site hematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All manuscripts should be submitted to the sponsor for review and comment prior to submission to the publisher.

DOCUMENTS (2):
  • Statistical Analysis Plan (2014-08-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT02274857/SAP_000.pdf
  • Study Protocol (2014-06-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT02274857/Prot_001.pdf